CLINICAL TRIAL: NCT07405359
Title: A Randomized Trial of Pulmonary Vein Isolation Alone Versus Pulmonary Vein Isolation Plus Posterior Wall and Superior Vena Cava Isolation With Pulsed Field Ablation for Treatment of Persistent Atrial Fibrillation
Brief Title: PVI Alone Versus PVI Plus PWI and SVCI With PFA
Acronym: PVI-PLUS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Edward Gerstenfeld, MD (Other)
Responsible Party: Sponsor-Investigator, Edward Gerstenfeld, MD, Professor, Medicine, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 25-44799
Record Dates: First submitted 2026-01-21; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Persistent Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- PVI alone (Active Comparator): Afib ablation: PVI only
  Interventions: Device: PFA; Procedure: Implantable loop recorder
- PVI + PWI + SVCI (Experimental): Afib ablation: PVI + PWI + SVCI
  Interventions: Procedure: AF Ablation: PVI + PWI + SVCI; Device: PFA; Procedure: Implantable loop recorder

INTERVENTIONS:
Procedure: AF Ablation: PVI + PWI + SVCI — Patients randomized to the 'PVI only' arm will be receiving an Afib ablation using PFA targeting the pulmonary veins for isolation (PVI). Following PVI, in those patients randomized to PVI+, PFA will also be used to isolate the left atrial posterior wall, and the superior vena cava.
  Arms: PVI + PWI + SVCI
Device: PFA — PFA is FDA-approved for PVI and PWI. SVCI using PFA will be done for investigational purposes.
Procedure: Implantable loop recorder — Implantation of implantable loop recorder during ablation procedure for continuous heart monitoring during follow up.

SUMMARY:
Catheter based ablation of atrial fibrillation (AF) is an established treatment modality for rhythm control of AF, with pulmonary vein isolation (PVI) being the cornerstone of this technique. While pulmonary vein triggers are the predominant arrhythmia mechanism in paroxysmal AF, development of additional atrial substrate contributes to maintenance of AF in persistent AF. This is likely to account for the lower rates of freedom from recurrent AF following ablation in patients with persistent AF. Various adjunctive empiric ablation strategies, such as left atrial posterior wall isolation (PWI), superior vena cava isolation (SVCI), linear ablation, and ablation of complex fractionated atrial electrograms have been studied to address this limitation of PVI alone.

While observational data supports the safety and feasibility of Posterior Wall Isolation (PWI) and Superior Vena Cava Isolation (SVCI) with PFA, the efficacy of these strategies with PFA has not been demonstrated in randomized controlled trials. Whether mapping prior to ablation (i.e. detecting scar) predicts if PW and SVC sites are effective in improving ablation outcome is unknown.

This study will test the hypothesis of whether empiric addition of PW and SVC isolation with PFA to PVI improves outcome (freedom from atrial tachyarrhythmia at 1-year). The investigators therefore propose a randomized controlled trial to compare the efficacy of Pulmonary Vein Isolation (PVI) alone versus PVI + PWI + SVCI in patients with persistent AF. The investigators hypothesize that the addition of PWI and SVCI to PVI in patients with persistent AF will provide improved freedom from AFIB off anti-arrhythmic drugs, without significantly increasing rates of procedural complications. Secondary analysis includes subgroups with posterior wall scar, procedure times, freedom from AFIB on or off anti arrhythmic drugs, etc.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years at their pre-procedure visit
* Persistent AF, defined as at least one continuous AF episode lasting at least seven days in duration, documented by a continuous monitor or 2 ECGs>7 days apart or ≥3 cardioversions
* Indicated and interested in ICM implant for monitoring post ablation
* Written informed consent obtained from subject and ability for subject to comply with the requirements of the study

Exclusion Criteria:

* Any prior atrial endocardial or epicardial ablation procedure, other than cavotricuspid isthmus ablation or supraventricular tachycardia
* Stroke or transient ischemic attack within the previous six months
* Gastrointestinal bleeding within the previous three months
* Implanted pacemaker or defibrillator
* Longstanding persistent AF (> 3 years)
* LA volume >80ml/m2
* Atrial septal occlusion device
* Current left atrial thrombus
* Left atrial appendage occlusion or closure device < 6 mos or with leak or prior DRT
* Mitral or Tricuspid valve clip or mechanical replacement or clip
* Hypertrophic cardiomyopathy
* Contraindication to femoral vascular access
* Congenital heart disease with residual anatomic abnormality
* Contraindication to, or unwillingness to use, systemic anticoagulation
* Pregnancy
* Left ventricular ejection fraction <30%
* Baseline creatinine >2.0 mg/dL
* Predicted life expectancy less than one year
* Refusal to receive ICM implant or allergy to ICM

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2026-02-14 (Estimated); Primary Completion 2028-08-14 (Estimated); Study Completion 2028-08-14 (Estimated)

PRIMARY OUTCOMES:
AF freedom | 12 months
  First recurrence of AT/AFL/AF > 1 hour after a 2-month blanking period Any 1) cardioversion 2) redo ablation or 3) escalation/change in AAD after the 2-month blanking period (allowing 3 months to stop AADs) is considered a failure of the primary endpoint

CONTACTS AND LOCATIONS:
Overall Officials: Edward Gerstenfeld, MD, MS, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No